CLINICAL TRIAL: NCT03869099
Title: To Document Pneumonia Case Management Practices in Selected Communities in Pakistan; A Qualitative Study
Brief Title: Pneumonia Case Management Practices in Pakistan
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: AC18006
Record Dates: First submitted 2018-11-26; First posted 2019-03-11 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pneumonia; Childhood Pneumonia; Infectious Disease; Acute Respiratory Infection
Keywords: Childhood pneumonia; acute respiratory illness; Pakistan
MeSH Terms: conditions — Pneumonia; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sindh
  Interventions: Other: Pneumonia Case Management Practices
- KPK
  Interventions: Other: Pneumonia Case Management Practices
- Punjab
  Interventions: Other: Pneumonia Case Management Practices
- Balochistan
  Interventions: Other: Pneumonia Case Management Practices

INTERVENTIONS:
Other: Pneumonia Case Management Practices — Standard practices of pneumonia case management at three levels of health care; community level, first level care facility and practitioner level, across Pakistan.

SUMMARY:
Pneumonia in Pakistan continues to be the leading killer of children under five. Although various national and provincial programs have tried to tackle this but they have not been able to achieve the desired outcomes. Additionally, there has been limited in depth evaluation of the practices of pneumonia management at various levels of the community. The investigators, therefore, aim to establish an understanding of pneumonia case management at three levels of healthcare - community, first level care facility and practitioner level. This will be conducted through observations of pneumonia case managements practices of healthcare providers at these three levels across the country by simulated patients. Observation checklists will be developed incorporating settings and behaviors. Observation sites will be randomly selected with 32 observations made in each province. The results of this study will yield the ground reality of pneumonia case management in Pakistan. Based on the results of this study, strategies can be devised to improve case management within the community with models of regular monitoring and supervision.

DETAILED DESCRIPTION:
Despite the availability of standard pneumonia management guidelines and multiple global efforts, pneumonia continues to be the leading killer of children under five, accounting to around 17% of the total under five deaths globally. It has been estimated that annually there are around 120 million episodes of pneumonia among children with around 14 million progressing to severe episodes. Out of these cases, close to 1.3 million children die with 81% of these deaths occurring in children under 2 years of age. Fifty two percent of these deaths occur in the Sub-Saharan region and South Asia with main contributions from India, Nigeria, Congo, Pakistan and Afghanistan. In Pakistan, pneumonia contributes to 16% of under-five mortality in the country having a well-defined yet poorly functional healthcare system.

Healthcare in Pakistan is provided through two sectors; public and private. The public sector includes community health workers, referred to as Lady Health Workers (LHWs) working under the National Program for Family planning and Primary Health Care. It also includes the First Level Care Facilities referred to as Basic Health Units (BHUs) and Rural Health Centres (RHCs) and district/tertiary care hospitals. The private sector includes the private clinic and private hospitals. The public sector provides healthcare free of cost or with minimal charges whereas the private sector is expensive as patients spend out-of-pocket for health service in this sector. This accounts to the wide difference of quality of care across both the sectors as the public sector is not funded adequately by the government to provide high quality services, due to only 2% of the Gross Domestic Product (GDP) assigned to healthcare. Irrespective of the public and private sector, case management of pneumonia in children under five is supposed to be followed uniformly across all sectors as training of the healthcare providers is standard across all cadres of care under various programs in the country. Despite that fact, the mortality and morbidity rate due to pneumonia in children under five remains unchanged in the country.

World Health Organization (WHO) and United Nations International Children's Emergency Fund (UNICEF) have developed multiple action/ intervention plans to curb pneumonia related morbidity and mortality in children under five and based on those plans Pakistan has launched multiple national programs. These programs include the National Acute Respiratory Illness (ARI) control program which was launched in 1989 with the main objectives of reducing severity and mortality due to pneumonia and rationalize the use of antimicrobials and other drugs for treatment of ARI. It was supported by WHO, UNICEF and United States Agency for International Development (USAID). While the program was ongoing, in 1990, in a National workshop on policy related research action plan, organized by the Ministry of Health, the Ministry of Planning and Development and the Aga Khan University (AKU), ARI was ranked sixth of fifteen priority areas for national policy-linked research. The National ARI Control program continued but WHO soon realized that this disease centric narrow approach has not been able to achieve its desired objectives. Therefore, it developed a more integrated approach and launched it globally as Integrated Management of Childhood Illnesses (IMCI) launched in Pakistan in 1998. The approach in IMCI focused on improving case management skills of health workers, strengthening the health system, and addressing family and community practices. Concerns were raised that this is yet another attempt to launch a child health intervention vertically. Duplicity was very much evident from the fact that ARI existed as an independent program and was also part of the IMCI package. Between 2004-2010, a USAID funded project called The Pakistan Initiative for Mothers and Newborns (PAIMAN) was undertaken which focused on improving the status of maternal and newborn health in 10 districts (19% of the national population), which later expanded to 24 districts across the four provinces and Azad Jammu and Kashmir in Pakistan. ARI was an important component in that project. The national Maternal, Neonatal and Child Health program (MNCH) was then launched in 2010 funded mainly by Development for International Development (DFID) implemented in 36 districts and ended after 5 years. It was focused on strengthening of management and organization mechanism of healthcare delivery systems. Under all these programs, selected health care professionals, both community and facility based, were trained on WHO standard of ARI case management. Looking at the unchanged mortality statistics, there is a concern that these trainings might have failed to change the case management practices within the community. It is perhaps due to the fact that the monitoring and evaluation was not a strong point of these programs.

There is limited data within Pakistan which reflects the status of the quality of current pneumonia case management practices throughout the three tiered health system (primary health facilities, secondary care hospitals, and tertiary care hospitals) as well as the private sector. There are a number of approaches which can be used to assess standard case management including recall based patient surveys, questionnaire surveys of knowledge, prescription/chart analysis and use of disguised patients to assess actual practice. A disguised patient is one who although suffers from a particular disease but acts as a disguised observer. Considering the use of disguised patients provides an actual picture of practice, therefore, it has been used extensively most recently. This process provides an assessment of the practitioners' knowledge of appropriate care and the actual care delivered, i.e., adherence to standard treatment guidelines. Such an approach in Pakistan can identify current pneumonia case management practices across the country because to-date no such study has been conducted in this field. The results of this study can help in informing design of future policies and interventions that can in turn assist in reducing pneumonia related morbidity and mortality.

Methodology:

This will be a qualitative study which will be conducted through participant observations over a period of 13 months across randomly selected sites in four provinces of Pakistan in addition to the federal capital. The provinces are Baluchistan, Khyber Pakhtunkhuwah (KPK), Punjab and Sindh.

After obtaining ethical clearance, an observation tool will be developed based on standard WHO guidelines and input from field experts. This tool will be pretested upon finalization. At the same time an advisory committee will also be formulated composed of expert pediatricians and public health professionals who will provide their input into the implementation protocol and the tool. Once the tool is finalized training will be conducted on the tool and then observations will be conducted.

Observation Sites:

Observations sites will be randomly selected from each of the four provinces and the capital through our specialized sampling software. Upon site selection, observations will be made across the following levels of healthcare: community level, first level care facility (FLCF) and practitioner level both in the public and private sector. The community level observations will include observation of the pneumonia case management by the Lady Health Workers (LHWs). LHWs are the primary care givers at the community level who cover around 60% of Pakistan. Their basic duties include education, counseling and basic management of the common maternal and child ailments. Each LHW covers around 100-120 household and visits each household once a month. The observations will be made either at the health house of the LHW or she will be requested to visit the household of the disguised patient.

The FLCF level will include observations made at the primary health care facilities which are the Basic Health Units (BHUs) and Rural Health Centres (RHCs). A basic health unit is located within a union council which is the smallest administrative unit in the Pakistani administrative system. Each basic health unit covers a catchment area of 25,000 households. Pakistan has around 5,290 Basic Health Units (BHUs) although not all are functional. Services provided at BHU are promotive, preventive, curative and referral. LHWs refer patients usually to BHUs. RHCs provide in-patient service as compared to BHUs. They usually have 10-20 beds and cover a catchment area of 100,000 people. The RHC provides promotive, preventive, curative, diagnostics and referral services apart from the in-patient services. It also provides clinical, logistical and managerial support to the BHUs, LHWs, and dispensaries that fall within its geographical limits. RHC also provides medico-legal, basic surgical, dental and ambulance services. There are around 552 RHCs in Pakistan.

The practitioner level observations will include those of practitioners at both the private and public sector. The public sector will include observations made in outpatient departments of selected tertiary care hospitals across the study sites. Observations made at the private practitioner level will include selected solitary private clinics or clinics within private hospitals. The community and FLCF level will represent practices within the rural community and the practitioner level will represent practices within the semi urban/urban communities.

Data Collectors:

A team of data collectors, who will be healthcare professionals, will be trained on appropriate administration of the observation tool upon recruitment. The training will also include an introduction to pneumonia, its signs and symptoms, diagnosis and management according to WHO guidelines. A 3 day interactive training workshop will be conducted whereby mock excesses will also be conducted. A total of three training will be conducted whereby data collectors from Islamabad (capital), Punjab and KPK will have one training as their participants can be managed to be brought in one location due to close proximity. Sindh and Baluchistan participants will have two separate trainings.

Recruitment of Patients' Caregiver and Conduction of Observations:

Each data collector will be provided a pre-defined list of addresses whereby the observations will be made. He/she will go to the location and will search the nearby community for cases of pneumonia in children under five. Once the cases have been identified, their caregivers will be sought. These caregivers are the primary individuals providing direct care to the child. Usually, these are the mothers, fathers, grandmothers or guardians of the child. They will explained the purpose of the study and will be requested to participate in the study to accompany the data collector who will be disguised as a relative/friend of the caregiver, to the health facilities and upon agreement will sign a consent form. This means that they will disguise as an acquaintance of the data collector who will take them to the healthcare professional to be observed. They will take the ill child along, give the history of that child to the healthcare professional and answer any relevant questions which will be asked by him/her and get the child examined and treated. In the meantime, the data collector will make the relevant observations based on the observation tool which will be filled after the visit. The data collector will not reveal that he/she is a healthcare professional. Additionally, the data collector will also take an audio recorder along to record the entire conversation which will help in filling up the observation tool later and also validate the visit. Once the visit is completed, the data collector will take the caregiver back to their premises and fill up the observation tool in tablets within one hour of the visit. Electronic Case Recruitment Forms (eCRFs) will be used for improved data quality, avoidance of manual data entry errors and confidentiality etc.

ELIGIBILITY:
Inclusion Criteria for Disguised Caretakers:

* Caregivers of children under five years of age. These are those individuals who provide direct care to the child. These could either be a mother, father, grandmother or guardian.
* The child under five under that caregiver's household must have symptoms of pneumonia/severe pneumonia
* Caregivers consenting to be a part of the study.

Exclusion Criteria for Disguised Caretakers:

• Caregivers of children under five suffering from co-morbidity with pneumonia.

Inclusion Criteria for Healthcare Professionals under Observation:

For LHWs:

* Those who have been practicing as LHWs for more than one year as identified by talking to the community.
* Those who belong to the catchment area of the selected study sites

For BHUs:

• Functional BHUs with at least one licensed healthcare provider.

For RHC:

• Functional RHCs with at least one licensed healthcare provider.

Public Practitioners:

* Paediatricians working in a government tertiary healthcare facility as a full time employee.
* In case the facility/location does not have specialist paediatricians, then general physicians working full time within that facility.

Private Practitioners:

* Full time/part time private paediatric practitioners working in either their private clinics or in private hospitals.
* In case the facility/location does not have specialist paediatricians, then general physicians working within that facility.

Exclusion Criteria for Healthcare Professionals under Observation:

• BHUs or RHCs run by non -licensed healthcare professionals as there are certain locations whereby due to lack of licensed healthcare professional's facility technicians tend to attend to the patients based on their experience.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Two data collectors per province will be recruited to make the observations making a total of 10 data collectors for all the locations. Additionally, one caregiver per observation will be recruited by the data collectors to accompany them. Meaning 160 caregivers will be recruited. This is to avoid inconvenience to the caregiver and their affected under five children. In case, a community is encountered whereby the cases of pneumonia are very few, then the same caregiver will be accompanied for observation of an LHW, BHU and RHC of that locality as these facilities are closely located. If despite this practice, number of observations are not achievable per site than an additional site will be provided to the data collector to visit.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
To assess number of healthcare providers providing standard pneumonia case management to under five children. | 13 months
  Standard case management practices regarding pediatric pneumonia comprising of components of history taking, examination, diagnosis and treatment across all provinces of Pakistan will be assessed. An observation checklist will be used to collect both qualitative and quantitative data. Quantitative data will be analyzed through descriptive and inferential statistics which will include province-wise reported frequencies of healthcare providers providing standard pneumonia case management to children under five. Whereas; qualitative data will be assessed through thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- MNCHRN, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03869099/Prot_SAP_000.pdf